CLINICAL TRIAL: NCT07043361
Title: Efficacy of Semaglutide in Glycemic Control, Weight Loss, and Improving Lipid Profile- the Role of Baseline Vitamin D Levels
Brief Title: Efficacy of Semaglutide in Glycemic Control, Weight Loss, and Improving Lipidogram- Role of Baseline Vitamin D Levels
Acronym: Semaglutide
Status: Completed | Type: Observational
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0034-23-LEU; Non applicable (Other Grant/Funding Number: Leumit health care system)
Record Dates: First submitted 2025-04-29; First posted 2025-06-29 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: Metabolic Disease
MeSH Terms: conditions — Metabolic Diseases | interventions — semaglutide

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- diabetic patients on semaglutide: we tested the relation between baseline vitamin D levels and metabolic amplification of semaglutide metabolic effects
  Interventions: Drug: semaglutide

INTERVENTIONS:
Drug: semaglutide — testing the effect of baseline vitamin D on metabolic effects of semaglutide

SUMMARY:
Objective: Semaglutide, a glucagon-like peptide-1 receptor agonist, is an established therapy for type 2 diabetes (T2D), offering robust glycemic control and weight reduction. Vitamin D has been implicated in metabolic regulation, yet its influence on semaglutide-induced outcomes remains unclear.

Research Design and Methods: the investigators conducted a cross-sectional analysis of 5,300 adults with T2D, enrolled in Leumit Health Services, who initiated semaglutide therapy between February 1, 2019, and December 31, 2022. All patients had documented serum 25-hydroxyvitamin D [25(OH)D] levels prior to treatment initiation. Metabolic outcomes- including glycemic control (HbA1c), body mass index (BMI), and lipid profile- were assessed at 12 months. Associations between baseline 25(OH)D levels and metabolic changes were evaluated using multivariable regression models, adjusted for demographic and clinical covariates.

DETAILED DESCRIPTION:
Semaglutide, a glucagon-like peptide-1 (GLP-1) receptor agonist, was initially approved for the treatment of type 2 diabetes mellitus (T2DM) due to its superior glucose-lowering efficacy compared to oral antidiabetic agents, with a favorable safety profile regarding hypoglycemia risk. In June 2021, the U.S. Food and Drug Administration (FDA) approved higher doses of semaglutide for long-term weight management, marking the first pharmacologic advancement in obesity treatment since 2014 (FDA, 2021).

Semaglutide exerts its effects through multiple mechanisms, including delayed gastric emptying, appetite suppression, enhanced glucose-stimulated insulin secretion from pancreatic β-cells, and reduced glucagon secretion. In individuals with overweight and obese, semaglutide induces substantial and sustained weight reduction, with an average decrease of approximately 14.9% of baseline body weight.

The pathophysiology of T2DM varies across racial and ethnic groups. For example, T2DM in Caucasian populations is primarily characterized by obesity and insulin resistance, whereas in East Asians, including the Japanese, early-onset β-cell dysfunction and insulin deficiency predominate. Consequently, the glycemic response to semaglutide is not uniform across populations. Notably, semaglutide predominantly enhances first-phase insulin secretion, an effect that may be particularly beneficial in individuals with insulin deficiency. Several blinded, controlled trials have demonstrated superior glycemic control with semaglutide in Asian populations, reinforcing the significance of insulin resistance versus insulin deficiency in determining its net metabolic effects.

While genetic and ethnic determinants of semaglutide response are largely non-modifiable, certain adjunctive interventions may optimize its therapeutic effects. Among these, vitamin D has emerged as a potential modulator of molecular pathways involved in metabolic regulation. In regard to diabetes control, vitamin D is a key immunomodulatory factor, and preclinical studies have demonstrated its protective effects against β-cell dysfunction in diabetes. In murine models, early vitamin D administration mitigated the inflammatory insults responsible for β-cell destruction, thereby preventing autoimmune diabetes onset. These findings are supported by human studies in prediabetic and newly diagnosed T2DM individuals, in whom long-term vitamin D supplementation (six months) significantly improved peripheral insulin sensitivity and β-cell function, potentially delaying diabetes progression.

Obesity has long been linked to vitamin D deficiency. While the role of vitamin D in weight loss remains debated, a recent meta-analysis highlighted its potential clinical efficacy in optimizing weight reduction. Specifically, three months of vitamin D supplementation in obese women significantly augmented weight loss and improved metabolic parameters.

Given the high prevalence of vitamin D deficiency, particularly among individuals with obesity and T2DM, supplementation may offer metabolic benefits.

To date, the relationship between vitamin D status and the metabolic effects of semaglutide has not been well characterized. In this retrospective cross-sectional study, The investigators aimed to investigate the association between baseline vitamin D levels and semaglutide-induced glycemic control and weight loss in an Israeli T2DM population.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes type II treated with semaglutide
* Available baseline vitamin D levels

Exclusion Criteria:

* Missing serum 25-hydroxyvitamin D (25[OH]D) data
* Pregnant or lactating females

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: diabetic patients on semaglutide treatment and with available baseline vitamin D levels
Sampling Method: Non-Probability Sample
Enrollment: 5300 (Actual)
Dates: Start 2023-12-18 (Actual); Primary Completion 2024-12-21 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
relative weight loss measured by BMI | 12 months from semaglutide initiation
  testing semaglutide induced weight loss as a function of baseline vitamin D levels
glycemic control using Hgb1C | 12 months from semaglutide initiation
  testing semaglutide induced glycemic control as a function of baseline vitamin D levels
lipid control using LDL and TG | 12 months from semaglutide initiation
  testing semaglutide induced lipid control as a function of baseline vitamin D levels

CONTACTS AND LOCATIONS:
Overall Officials: rami abo fanne, MD PhD, Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Leumit Health ccare system, Hadera, Israel

IPD SHARING:
Plan to Share IPD: No
data is personal and secured

REFERENCES:
- [Background] Miles KE, Kerr JL. Semaglutide for the Treatment of Type 2 Diabetes Mellitus. J Pharm Technol. 2018 Dec;34(6):281-289. doi: 10.1177/8755122518790925. Epub 2018 Jul 30. PMID 34861016
- [Background] Andersen A, Knop FK, Vilsboll T. A Pharmacological and Clinical Overview of Oral Semaglutide for the Treatment of Type 2 Diabetes. Drugs. 2021 Jun;81(9):1003-1030. doi: 10.1007/s40265-021-01499-w. Epub 2021 May 8. PMID 33964002
- [Background] Davies MJ, Aroda VR, Collins BS, Gabbay RA, Green J, Maruthur NM, Rosas SE, Del Prato S, Mathieu C, Mingrone G, Rossing P, Tankova T, Tsapas A, Buse JB. Management of hyperglycaemia in type 2 diabetes, 2022. A consensus report by the American Diabetes Association (ADA) and the European Association for the Study of Diabetes (EASD). Diabetologia. 2022 Dec;65(12):1925-1966. doi: 10.1007/s00125-022-05787-2. Epub 2022 Sep 24. PMID 36151309
- [Background] Evans M, Morgan AR, Bain SC, Davies S, Hicks D, Brown P, Yousef Z, Dashora U, Viljoen A, Beba H, Strain WD. Meeting the Challenge of Virtual Diabetes Care: A Consensus Viewpoint on the Positioning and Value of Oral Semaglutide in Routine Clinical Practice. Diabetes Ther. 2022 Feb;13(2):225-240. doi: 10.1007/s13300-021-01201-z. Epub 2022 Jan 19. PMID 35044569
- [Background] Kalra S, Kapoor N. Oral Semaglutide: Dosage in Special Situations. Diabetes Ther. 2022 Jun;13(6):1133-1137. doi: 10.1007/s13300-022-01265-5. Epub 2022 May 7. PMID 35532859
- [Background] Wilding JPH, Batterham RL, Calanna S, Davies M, Van Gaal LF, Lingvay I, McGowan BM, Rosenstock J, Tran MTD, Wadden TA, Wharton S, Yokote K, Zeuthen N, Kushner RF; STEP 1 Study Group. Once-Weekly Semaglutide in Adults with Overweight or Obesity. N Engl J Med. 2021 Mar 18;384(11):989-1002. doi: 10.1056/NEJMoa2032183. Epub 2021 Feb 10. PMID 33567185
- [Background] Seino Y, Kuwata H, Yabe D. Incretin-based drugs for type 2 diabetes: Focus on East Asian perspectives. J Diabetes Investig. 2016 Apr;7 Suppl 1(Suppl 1):102-9. doi: 10.1111/jdi.12490. Epub 2016 Apr 18. PMID 27186364
- [Background] Yabe D, Seino Y, Fukushima M, Seino S. beta cell dysfunction versus insulin resistance in the pathogenesis of type 2 diabetes in East Asians. Curr Diab Rep. 2015 Jun;15(6):602. doi: 10.1007/s11892-015-0602-9. PMID 25944304
- [Background] Kakei M, Yoshida M, Dezaki K, Ito K, Yamada H, Funazaki S, Kawakami M, Sugawara H, Yada T. Glucose and GTP-binding protein-coupled receptor cooperatively regulate transient receptor potential-channels to stimulate insulin secretion [Review]. Endocr J. 2016 Oct 29;63(10):867-876. doi: 10.1507/endocrj.EJ16-0262. Epub 2016 Jul 17. PMID 27321586
- [Background] Yosida M, Dezaki K, Uchida K, Kodera S, Lam NV, Ito K, Rita RS, Yamada H, Shimomura K, Ishikawa SE, Sugawara H, Kawakami M, Tominaga M, Yada T, Kakei M. Involvement of cAMP/EPAC/TRPM2 activation in glucose- and incretin-induced insulin secretion. Diabetes. 2014 Oct;63(10):3394-403. doi: 10.2337/db13-1868. Epub 2014 May 13. PMID 24824430
- [Background] Yabe D, Yamada Y, Kaku K, Nishida T, Sato T, Seino Y. Efficacy and safety of once-weekly semaglutide in Japanese individuals with type 2 diabetes by baseline age and body mass index. J Diabetes Investig. 2022 Jul;13(7):1161-1174. doi: 10.1111/jdi.13773. Epub 2022 Mar 9. PMID 35174649
- [Background] Kim YG, Hahn S, Oh TJ, Park KS, Cho YM. Differences in the HbA1c-lowering efficacy of glucagon-like peptide-1 analogues between Asians and non-Asians: a systematic review and meta-analysis. Diabetes Obes Metab. 2014 Oct;16(10):900-9. doi: 10.1111/dom.12293. Epub 2014 Apr 15. PMID 24655583
- [Background] Kang YM, Cho YK, Lee J, Lee SE, Lee WJ, Park JY, Kim YJ, Jung CH, Nauck MA. Asian Subpopulations May Exhibit Greater Cardiovascular Benefit from Long-Acting Glucagon-Like Peptide 1 Receptor Agonists: A Meta-Analysis of Cardiovascular Outcome Trials. Diabetes Metab J. 2019 Aug;43(4):410-421. doi: 10.4093/dmj.2018.0070. Epub 2018 Dec 27. PMID 30604598
- [Background] Gysemans CA, Cardozo AK, Callewaert H, Giulietti A, Hulshagen L, Bouillon R, Eizirik DL, Mathieu C. 1,25-Dihydroxyvitamin D3 modulates expression of chemokines and cytokines in pancreatic islets: implications for prevention of diabetes in nonobese diabetic mice. Endocrinology. 2005 Apr;146(4):1956-64. doi: 10.1210/en.2004-1322. Epub 2005 Jan 6. PMID 15637289
- [Background] Lemieux P, Weisnagel SJ, Caron AZ, Julien AS, Morisset AS, Carreau AM, Poirier J, Tchernof A, Robitaille J, Bergeron J, Marette A, Vohl MC, Gagnon C. Effects of 6-month vitamin D supplementation on insulin sensitivity and secretion: a randomised, placebo-controlled trial. Eur J Endocrinol. 2019 Sep;181(3):287-299. doi: 10.1530/EJE-19-0156. PMID 31344685
- [Background] Perna S. Is Vitamin D Supplementation Useful for Weight Loss Programs? A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Medicina (Kaunas). 2019 Jul 12;55(7):368. doi: 10.3390/medicina55070368. PMID 31336940
- [Background] Subih HS, Zueter Z, Obeidat BM, Al-Qudah MA, Janakat S, Hammoh F, Sharkas G, Bawadi HA. A high weekly dose of cholecalciferol and calcium supplement enhances weight loss and improves health biomarkers in obese women. Nutr Res. 2018 Nov;59:53-64. doi: 10.1016/j.nutres.2018.07.011. Epub 2018 Jul 25. PMID 30442233

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-18): https://cdn.clinicaltrials.gov/large-docs/61/NCT07043361/Prot_SAP_001.pdf